CLINICAL TRIAL: NCT03099486
Title: A Pilot Phase II, Single Arm, Open Label, Investigator-initiated Clinical Trial of Regorafenib Plus 5-Fluorouracil/Leucovorin (5FU/LV) Beyond Progression on Regorafenib Monotherapy in Metastatic Colorectal Cancer (mCRC)
Brief Title: Regorafenib Plus 5-Fluorouracil/Leucovorin Beyond Progression in mCRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative change
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1023; GI-094 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2017-03-23; First posted 2017-04-04 (Actual); Results first posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regorafenib + 5FU/LV Treatment Arm (Experimental)
  Interventions: Drug: Regorafenib; Drug: 5-FU; Drug: Leucovorin

INTERVENTIONS:
Drug: Regorafenib — The dose of Regorafenib is 160 mg PO daily D1-D21 of 28-day cycle or last tolerated dose while on Regorafenib monotherapy.
Drug: 5-FU — 5-FU dose D1 and D15 of 28 day cycle i400 mg/m2 bolus over 10 mins followed by 2400 mg/m2 continuous infusion over 46 hours
Drug: Leucovorin — D1 and D15 of 28 day cycle Leucovorin 400 mg/m2 over 2 hours,

SUMMARY:
This is a single arm open label pilot phase II trial of Regorafenib PO plus 5-FU/LV infusion in 15 mCRC patients who progressed on prior Regorafenib monotherapy as well as 5-FU containing chemotherapy combinations.The study will enroll mCRC patients with prior progression on standard multi-agent combination chemotherapy and progression on regorafenib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. mCRC with prior progression on standard multi-agent combination chemotherapy and regorafenib as a standard approved monotherapy. Progression on prior regorafenib is required for inclusion in this clinical study. Prior regimens may include FOLFOX -/+ bevacizumab, FOLFIRI -/+ bevacizumab or -/+ cetuximab (if KRAS wild-type) or panitumumab (if KRAS wilt-type). Other prior regimens may include 5-FU or capecitabine -/+ bevacizumab, irinotecan -/+ cetuximab or panitumumab, FOLFIRI -/+ ziv-aflibercept or ramucirumab.
2. Patients treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy. Patients who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated. Patients who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed in the study.
3. Patients previously treated with chemotherapy must have at least 4 weeks period between the last dose of previous chemotherapy and the first dose in this clinical study. Patients previously treated with biologics such as Avastin, Zaltrap, Erbitux, and Vectibix must have at least 6 weeks period between the last dose of previous chemotherapy and the first dose in this clinical study.
4. Measurable metastatic disease that is refractory.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. Patients are included regardless of KRAS/NRAS, BRAF, p53, or microsatellite instability (MSI) status
7. Age ≥ 18 years.
8. Life expectancy of at least 8 weeks (2 months).
9. Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
10. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

    * Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
    * Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
    * Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
    * Serum creatinine ≤ 1.5 x the ULN
    * International normalized ratio (INR)/ Partial thromboplastin time (PTT) ≤ 1.5 x ULN.
    * Platelet count > 100000 /mm3, hemoglobin (Hb) > 9 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm3. Blood transfusion to meet the inclusion criteria will not be allowed.
11. Subject must be able to swallow and retain oral medication.
12. Up to 5 of the 15 patients will be allowed to have had other approved or investigational drugs after prior progression of Regorafenib monotherapy. (all patients enrolled in this trial must have had prior progression on regorafenib therapy). This may include TAS102, off-label therapy that may have been prescribed based on tumor genomic profiling or any investigational agents on a clinical trial.
13. No more than grade 2 toxicity with last previous cycle of regorafenib mono therapy.

Exclusion Criteria:

1. Patients receiving any concurrent investigational agents
2. Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
3. Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management.
4. Active or clinically significant cardiac disease including:

   * Congestive heart failure - New York Heart Association (NYHA) > Class II.
   * Active coronary artery disease.
   * Suspected Long QT syndrome defined as QTc interval > 500 milliseconds at baseline.
   * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
   * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
5. Evidence or history of bleeding diathesis or coagulopathy.
6. Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
7. Subjects diagnosed with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 3 months of start of study treatment.
8. Patients with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated nonmelanoma skin carcinoma, noninvasive aerodigestive neoplasms, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed; all cancer treatments must be completed at least 3 years prior to registration.
9. Patients with phaeochromocytoma.
10. Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
11. Ongoing infection > Grade 2 NCI-CTCAE v4.0.
12. Symptomatic metastatic brain or meningeal tumors.
13. Presence of a non-healing wound, non-healing ulcer, or bone fracture.
14. Major surgical procedure or significant traumatic injury within 28 days before start of study medication
15. Renal failure requiring hemo-or peritoneal dialysis.
16. Dehydration Grade ≥1 NCI-CTCAE v4.0.
17. Patients with seizure disorder requiring medication.
18. Persistent proteinuria ≥ Grade 3 per NCI-CTCAE v4.0 (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
19. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
20. Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.0 Grade 2 dyspnea).
21. History of organ allograft (including corneal transplant).
22. Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
23. Any malabsorption condition.
24. Women who are pregnant or breast-feeding.
25. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
26. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
27. Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin) or with heparins and heparinoids.

    a. However, prophylactic anticoagulation as described below is allowed: i. Low dose warfarin (1 mg orally, once daily) with PT-INR ≤ 1.5 x ULN is permitted.

    ii. Low dose aspirin (≤ 100 mg daily). iii. Prophylactic doses of heparin. iv. Low molecular weight heparin Subjects who are prophylactically treated with an agent such as warfarin or heparin require close monitoring (day5 of cycle 1 and day 1 of each cycle) of their INR/PTT. If either of these values are above the therapeutic range, the doses should be modified and the assessments should be repeated weekly until they are stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Namrata Vijayvergia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 1
  Black or African American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 2 Months
Description: PFS at 2 months in mCRC patients who progress on regorafenib monotherapy and are treated with regorafenib and 5-FU/LV combination therapy.
Time Frame: 2 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
Number analyzed (Participants) | 2
months | NA [NA to NA] — Study was halted prematurely due to low accrual, not enough data obtained for analysis.

2. Secondary Outcome: Overall Survival Rate
Description: Overall survival will be calculated from the day of first treatment until death
Time Frame: 1 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
Number analyzed (Participants) | 2
months | NA [NA to NA] — Study was halted prematurely due to low accrual, not enough data obtained for analysis.

3. Secondary Outcome: Best Overall Response
Description: This will be calculated from the day of first treatment dose until disease progression or death, whichever occurs earlier
Time Frame: 1-2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
Number analyzed (Participants) | 2
Participants | NA — Study was halted prematurely due to low accrual, not enough data obtained for analysis.

4. Secondary Outcome: Number of Toxicities Due to Regorafenib and 5-FU/LV Combination Therapy
Description: Number of toxicities due to combination therapy will be summarized by frequencies and grades of toxicities due to the combination therapy according to CTCAE 4.03 criteria
Time Frame: 1-2 years
Measure: Number (95% Confidence Interval); unit: toxicities
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
Number analyzed (Participants) | 2
toxicities | NA [NA to NA] — Study was halted prematurely due to low accrual, not enough data obtained for analysis.

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Regorafenib + 5FU/LV Treatment Arm
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib + 5FU/LV Treatment Arm (N=2)
Moderate Congestive Heart Failure (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib + 5FU/LV Treatment Arm (N=2)
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Chills (General disorders) | 1
Edema Limbs (General disorders) | 1
Fever (General disorders) | 1
Pain (General disorders) | 1
Infection (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Weight Loss (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 1
Platelet Count Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarsness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Heart Failure (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Agitation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03099486/Prot_SAP_001.pdf
  • Informed Consent Form (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT03099486/ICF_000.pdf